CLINICAL TRIAL: NCT06842381
Title: Electrotherapy Combined With Neck Exercises for Non-Specific Neck Pain: Telerehabilitation Versus Face-to-Face Program: Study Protocol for a Multicenter Randomized Controlled Trial
Brief Title: Electrotherapy Combined With Neck Exercises for Non-Specific Neck Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adelaida María Castro-Sánchez (Other)
Collaborators: Andaluz Health Service (Other Government)
Responsible Party: Sponsor-Investigator, Adelaida María Castro-Sánchez, Full Professor, Universidad de Almeria
Organization: Universidad de Almeria (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SICEIA-2024-000820
Record Dates: First submitted 2025-02-12; First posted 2025-02-24 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Program (Experimental): Patients will be instructed in the therapeutic approach through a telerehabilitation program using a portable TENS (Transcutaneous Electrical Nerve Stimulation) with a specific program for cervical pain (ENRAF NONIOUS Iberica, SA, Spain) while performing McKenzie exercises. The specific program will consist of a conventional low-frequency, high-phase duration TENS (80 Hz/200 μs) applied directly to the cervical area using four electrodes (5x5 cm) at the bilateral paravertebral level. In patients who present radicular pain, the electrodes will be placed along the path of the affected nerve.
  Interventions: Other: Face to Face Program
- Face to Face Program (Active Comparator): Patients will be instructed in the therapeutic approach through a face to face program using a portable TENS (Transcutaneous Electrical Nerve Stimulation) with a specific program for cervical pain (ENRAF NONIOUS Iberica, SA, Spain) while performing McKenzie exercises. The specific program will consist of a conventional low-frequency, high-phase duration TENS (80 Hz/200 μs) applied directly to the cervical area using four electrodes (5x5 cm) at the bilateral paravertebral level. In patients who present radicular pain, the electrodes will be placed along the path of the affected nerve.
  Interventions: Other: Telerehabilitation Program

INTERVENTIONS:
Other: Telerehabilitation Program — A support system for the treatment of cervical pain based on Web technologies will be used, accredited as a health website. This system has a structure based on 4 sections: database treatment, database user profiles, recommendations, and feedback/biofeedback procedures. This system allows the registration and introduction of a subject, and modification of a treatment with electroanalgesia and exercises, according to the symptomatic evolution of the pain. It is based on an initial patient assessment system.
  Arms: Face to Face Program
Other: Face to Face Program — Electroanalgesia therapy and the McKenzie exercise protocol will be applied by six therapists with more than 10 years of experience in both procedures. This program will be developed in the Health Sciences clinical units of the Universities of Almeria, Granada and Malaga.
  Arms: Telerehabilitation Program

SUMMARY:
Objectives: The objective of this study is to compare the effectiveness of telerehabilitation versus a face-to-face program in the therapeutic approach to non-specific neck pain through exercise and analgesic electrotherapy.

Methods: Randomized clinical trial on 100 participants with nonspecific neck pain who will be randomized into two groups to receive analgesic electrotherapy combined with a cervical exercise program through telemedicine or face to face. A total of 24 sessions will be applied over 8 weeks. Demographic and clinical data, disability, pain intensity, kinesiophobia, isometric spinal muscle strength, quality of life, and cervical mobility will be collected. Assessments will be performed at the beginning of the study (baseline), at 8 weeks (post-treatment) and 2 months after the end of the intervention (follow-up).

DETAILED DESCRIPTION:
Introduction: Neck pain is a common problem in the working-age population, with a high recurrence rate and one of the highest health costs globally. Exercise is considered one of the keys in the management of this pathology, and electrotherapy is consolidated as a safe and proven analgesic measure. Telemedicine facilitates access to health care by eliminating geographical barriers and reducing costs, allowing consultations from any location and favoring the patient's work-life balance. The widespread availability of smartphones, tablets and computers makes telerehabilitation more accessible than ever.

Objectives: The objective of this study is to compare the effectiveness of telerehabilitation versus a face-to-face program in the therapeutic approach to non-specific neck pain through exercise and analgesic electrotherapy.

Methods: Randomized clinical trial with 100 participants with non-specific neck pain who will be randomized into two groups to receive analgesic electrotherapy combined with a cervical exercise program through telemedicine or face to face. A total of 24 sessions will be applied over 8 weeks. Demographic and clinical data, disability, pain intensity, kinesiophobia, isometric spinal muscle strength, quality of life, and cervical mobility will be collected. Assessments will be performed at the beginning of the study (baseline), at 8 weeks (post-treatment) and 2 months after the end of the intervention (follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between the ages of 30 and 65, with a medical diagnosis of cervical pain of non-specific origin,

  * Acceptance and signature of informed consent for voluntary participation in the research study.
  * Not receiving physical therapy.
* Chronic cervical pain lasting 3 months or more and not receiving any other type of physiotherapy treatment.

Exclusion Criteria:

* Patients undergoing rehabilitation treatment for pathologies of cervical origin.
* Patients have osteosynthesis material at the cervical level and/or cardiac complications, epilepsy or tumors.
* Patients who have undergone radiotherapy in the last 6 months.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Neck disability index | At baseline, 8 weeks and 6 months (follow up).
  The neck disability index consists of 10 questions addressing functional activities such as personal care, lifting, reading, work, driving, sleeping, recreational, pain intensity, concentration and headache. Each item will be scored on a scale from 0 (no limitation). (severe limitation or inability to perform the activity). The total score will be calculated by summing the item scores, dividing by the maximum possible score of 50 (if all 10 questions are answered), and multiplying by 100 to generate a percentage. A score of 0% indicates full independence, while 100% represents complete dependence.

SECONDARY OUTCOMES:
Pain (Visual Analog Scale) | At baseline, 8 weeks and 6 months (follow up).
  Pain will be assessed with the Visual Analog Scale (VAS), which assesses the pain intensity and degree of relief experienced by the patient (scored of 0 = no pain; 10 = unbearable pain).
McGill Pain Questionnaire (Disability) | At baseline, 8 weeks and 6 months (follow up).
  The McGill Pain Questionnaire is a self-reporting measure of pain used for patients with a number of diagnoses. It assesses both quality and intensity of subjective pain. The MPQ is a multi-dimesional tool for pain assessment and it has three components, which are the sensory intensity, the cognitive evaluation of pain and the emotional impact of pain. Interpretation: • minimum pain score: 0 (would not be seen in a person with true pain). • maximum pain score: 78. • The higher the pain score the greater the pain.
Quality of Life (SF-36 quality of life questionnaire) | At baseline, 8 weeks and 6 months (follow up).
  The SF-36 quality of life questionnaire assesses 8 domains including physical functioning, physical role, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Scores range from 0 to 100% (with higher scores indicating greater health), reflecting the individual's self-perceived health-related quality of life.
Quality of Sleep (Pittsburgh Quality of Sleep Questionnaire Index) | At baseline, 8 weeks and 6 months (follow up).
  The Pittsburgh Quality of Sleep Questionnaire Index (PSQI) will be used to study the quality of sleep. It comprises 24 items where the subjects respond to 19 of these items, and individual living in the same dwelling (or hospital room) responds to the remaining 5. Scores are obtained on each of 7 components of sleep quality: subjective quality, sleep latency, sleep duration, habitual sleep efficacy, sleep perturbations, use of hypnotic medication, and daily dysfunction. Using a four-point, Likert-type scale, respondents indicate how frequently they exhibit certain sleep behaviors (0 = "few," 1 = "sometimes," 2 = "often," and 3 = "almost always"). Scores on items belong to factors 2 and 5 (restoration after sleep and satisfaction with sleep) and are reversed before being tallied. Total scores can range from 0 to 84, with higher scores demoting more acute sleep problems.
Tampa scale for kinesiophobia | At baseline, 8 weeks and 6 months (follow up).
  The 17-item Tampa scale for kinesiophobia assesses fear of movement or of injury or reinjury. Participants rate their beliefs regarding kinesiophobia on a 4-point Likert scale, ranging from "strongly disagree" to "strongly agree".
Pain Catastrophizing Scale | At baseline, 8 weeks and 6 months (follow up).
  The Pain Catastrophizing Scale (PCS) is a self-assessment questionnaire to examine catastrophizing in clinical and nonclinical populations. Catastrophizing is commonly described as an exaggerated negative orientation toward noxious stimuli and plays an important role in experiencing and coping with pain. The PCS consists of 13 statements containing a number of thoughts and feelings one may experience when having pain. The items are divided into the categories of rumination, magnification and helplessness, with each item scored on a 5-point scale. The PCS consists of 13 statements containing several thoughts and feelings one may experience when having pain.
Cervical Range of Motion (Pro Motion Capture. Werium) | At baseline, 8 weeks and 6 months (follow up).
  Cervical range of motion is assessed with the patient sitting comfortably on a chair, with both feet flat on the floor, hips and knees at 90º of flexion, and buttocks positioned against the back of the chair.
Spinal Isometric Strength (SIS) | At baseline, 8 weeks and 6 months (follow up).
  The investigators will measure the maximum isometric strength of the neck extensor muscles using a hand-held dynamometer (HHD). The patient will remain seated in a chair, with their feet flat on the floor, their hips and knees at 90º of flexion and the neck in the anatomical position, the patient will hold the HHD with both hands resting on their occiput, opposing the extension, and will be asked to perform a progressive isometric cervical extension for 3 seconds until reaching their maximum level of strength.
Neck Flexor Muscle Endurance Test (NFME) | At baseline, 8 weeks and 6 months (follow up).
  To measure the isometric endurance of the neck flexors, the investigators will place the patient in a supine position and ask him/her to perform a double chin tuck, which he/she must maintain throughout the test. While maintaining this position, he/she must flex his/her neck until his/her head is 2.5 cm off the table and maintain this position for as long as possible. The evaluator will time the duration of the test, which will be terminated if the patient loses the position for more than one second or asks to end due to fatigue or pain.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Almeria, Almería, Almeria, Spain

IPD SHARING:
Plan to Share IPD: Yes
The study data will be available by email at adelaid@ual.es, provided that a reasonable request is made with justification for its scientific use and that citation is guaranteed.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning with the first article publication; ending 5 years following article publication.
Access Criteria: Data will be accessed via the contact email adelaid@ual.es, provided that its scientific use and citation of our protocol are guaranteed.
  Access provided at no cost, unless repository policies require otherwise.

REFERENCES:
- [Result] Ozden F, Sari Z, Karaman ON, Aydogmus H. The effect of video exercise-based telerehabilitation on clinical outcomes, expectation, satisfaction, and motivation in patients with chronic low back pain. Ir J Med Sci. 2022 Jun;191(3):1229-1239. doi: 10.1007/s11845-021-02727-8. Epub 2021 Aug 6. PMID 34357527
- [Result] Hinman RS, Campbell PK, Kimp AJ, Russell T, Foster NE, Kasza J, Harris A, Bennell KL. Telerehabilitation consultations with a physiotherapist for chronic knee pain versus in-person consultations in Australia: the PEAK non-inferiority randomised controlled trial. Lancet. 2024 Mar 30;403(10433):1267-1278. doi: 10.1016/S0140-6736(23)02630-2. Epub 2024 Mar 7. PMID 38461844
- [Result] Xiang W, Wang JY, Ji BJ, Li LJ, Xiang H. Effectiveness of Different Telerehabilitation Strategies on Pain and Physical Function in Patients With Knee Osteoarthritis: Systematic Review and Meta-Analysis. J Med Internet Res. 2023 Dec 4;25:e40735. doi: 10.2196/40735. PMID 37982411
- [Result] Lara-Palomo IC, Gil-Martinez E, Ramirez-Garcia JD, Capel-Alcaraz AM, Garcia-Lopez H, Castro-Sanchez AM, Antequera-Soler E. Efficacy of e-Health Interventions in Patients with Chronic Low-Back Pain: A Systematic Review with Meta-Analysis. Telemed J E Health. 2022 Dec;28(12):1734-1752. doi: 10.1089/tmj.2021.0599. Epub 2022 May 9. PMID 35532971
- [Result] Villatoro-Luque FJ, Rodriguez-Almagro D, Aibar-Almazan A, Fernandez-Carnero S, Pecos-Martin D, Ibanez-Vera AJ, Castro-Martin E, Achalandabaso-Ochoa A. Telerehabilitation for the treatment in chronic low back pain: A randomized controlled trial. J Telemed Telecare. 2025 Jun;31(5):637-646. doi: 10.1177/1357633X231195091. Epub 2023 Aug 30. PMID 37649362
- [Result] Janela D, Costa F, Molinos M, Moulder RG, Lains J, Francisco GE, Bento V, Cohen SP, Correia FD. Asynchronous and Tailored Digital Rehabilitation of Chronic Shoulder Pain: A Prospective Longitudinal Cohort Study. J Pain Res. 2022 Jan 8;15:53-66. doi: 10.2147/JPR.S343308. eCollection 2022. PMID 35035234
- [Result] Bobos P, Pereira TV, Pouliopoulou DV, Charakopoulou-Travlou M, Nazari G, MacDermid JC. Which Remote Rehabilitation Interventions Work Best for Chronic Musculoskeletal Pain and Depression? A Bayesian Network Meta-Analysis. J Orthop Sports Phys Ther. 2024 Jun;54(6):361-376. doi: 10.2519/jospt.2024.12216. PMID 38406873
- [Result] Sivertsson J, Sernert N, Ahlund K. Exercise-based telerehabilitation in chronic low back pain - a scoping review. BMC Musculoskelet Disord. 2024 Nov 23;25(1):948. doi: 10.1186/s12891-024-07952-7. PMID 39580408
- [Result] Peterson G, Peolsson A. Efficacy of Neck-Specific Exercise With Internet Support Versus Neck-Specific Exercise at a Physiotherapy Clinic in Chronic Whiplash-Associated Disorders: Multicenter Randomized Controlled Noninferiority Trial. J Med Internet Res. 2023 Jun 20;25:e43888. doi: 10.2196/43888. PMID 37338972
- [Result] Nanda U, Luo J, Wonders Q, Pangarkar S. Telerehabilitation for Pain Management. Phys Med Rehabil Clin N Am. 2021 May;32(2):355-372. doi: 10.1016/j.pmr.2021.01.002. Epub 2021 Mar 6. PMID 33814062
- [Result] Cuenca-Martinez F, Lopez-Bueno L, Suso-Marti L, Varangot-Reille C, Calatayud J, Herranz-Gomez A, Romero-Palau M, Casana J. Implementation of Online Behavior Modification Techniques in the Management of Chronic Musculoskeletal Pain: A Systematic Review and Meta-Analysis. J Clin Med. 2022 Mar 24;11(7):1806. doi: 10.3390/jcm11071806. PMID 35407414